CLINICAL TRIAL: NCT01217476
Title: A Phase III, Double-Blind, Placebo Controlled, Parallel Group, International, Multicenter Study of 12 Weeks Treatment With Trafermin 0.01% Spray in Patients With Diabetic Foot Ulcer of Neuropathic Origin
Brief Title: The TRAfermin in Neuropathic Diabetic Foot Ulcer Study - Northern Europe The TRANS-North Study
Acronym: TRANS-North
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Olympus Biotech Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TFM-CL3-002; 2010-021015-16 (EudraCT Number)
Record Dates: First submitted 2010-10-07; First posted 2010-10-08 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-08

CONDITIONS: Diabetic Foot Ulcer of Neuropathic Origin
Keywords: Diabetic foot; Neuropathic; Wound; Growth factor
MeSH Terms: conditions — Diabetic Foot; Wounds and Injuries | interventions — trafermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trafermin 0.01% spray (Active Comparator)
  Interventions: Drug: Trafermin 0.01% spray
- Matching placebo spray (Placebo Comparator)
  Interventions: Drug: Trafermin 0.01% spray

INTERVENTIONS:
Drug: Trafermin 0.01% spray — For ulcers with a maximum diameter (longest axis) of less or equal to 6 cm, the daily dose of trafermin 0.01% spray is 5 puffs (30 microgram) sprayed onto the wound surface. If the maximum diameter (longest axis) of the ulcer is >6 cm, the ulcer should be sprayed in two parts, i.e. 5 puffs (30 microgram) sprayed onto each half of the wound surface

SUMMARY:
Trafermin is a recombinant human basic fibroblast growth factor (bFGF; original development code, KCB-1), which is manufactured by genetic engineering using Escherichia coli by Kaken Pharmaceutical Co., Ltd. (Tokyo, Japan). Trafermin 0.01% cutaneous spray product kit consisting of a glass bottle containing lyophilized trafermin, a glass bottle with solvent for solution and a spray part to fit the glass bottle after reconstitution of the final product.

We conduct a multinational, randomized, double-blind, placebo controlled, parallel-group, multicentre study consisting of a placebo run-in phase (2w), a treatment phase (max. 12w) and a follow-up phase (3mo+6mo). The primary objective of the study is to demonstrate a superior wound closure rate of diabetic foot ulcers (DFUs) of neuropathic origin after a maximum of 12 weeks topical daily application of trafermin 0.01% spray compared with placebo, in addition to best local care (off-loading, dressings). Approximately 210 patients will be randomized and it is planned that this study will be conducted at approximately 40 investigational sites in Europe.

ELIGIBILITY:
Selection Criteria

Patients who fulfill all of the following criteria (and none of the exclusion criteria described below) are eligible to enter the placebo run-in phase of the study:

1. Provide written informed consent to participate.
2. Male or female patients age 18 years or older.
3. Type 1 or 2 diabetes.
4. A single full-thickness DFU that has been present for at least 2 weeks.
5. DFU wound surface area below or equal 34 cm2 on the target foot.
6. No exposure of bone in the target DFU.
7. Neuropathy confirmed by loss of protective sensation to monofilament test (Semmes-Weinstein 5.07 monofilament).
8. No predominant ischemia requiring further exploration or treatment, and confirmed by either:

   * ABPI on the target leg (>0.9; below or equal 1.3) or if ABPI is >1.3 or is not assessable,TBPI on target foot ³above or equal 0.7, OR
   * ABPI on target leg (above or equal 0.7 - below or equal 0.9) or if ABPI is >1.3 or is not assessable, TBPI on target foot <0.7, AND a toe blood pressure >40 mmHg

Inclusion Criteria

Patients who fulfill all of the following criteria are eligible for randomization:

1. All of the selection criteria and none of the exclusion criteria are met.
2. Completed the 2-week placebo run-in period during which they were compliant to off-loading and to daily application of placebo spray, without major protocol violation. Compliance with the placebo run-in treatment regimen must be "excellent" or "acceptable".
3. Glycosylated hemoglobin (HbA1c) below or equal 10% (from a blood sample taken during the placebo run-in period).
4. Non-infected target foot DFU of confirmed neuropathic origin with:

   * ABPI on the target leg (>0.9; below or equal 1.3) or if ABPI is >1.3 or is not assessable, TBPI on target foot above or equal 0.7, OR
   * ABPI on target leg (above or equal 0.7 - below or equal 0.9) or if ABPI is >1.3 or is not assessable, TBPI on target foot <0.7, AND a toe blood pressure >40 mmHg
5. Target DFU appropriately debrided (<10% black and at least 50% of red/pink on a colorimetric scale)
6. Target DFU of grade A1 or A2 on the University of Texas Wound Classification System or of Grade 1 or 2 of the Wagner classification.
7. DFU surface area between above or equal 0.9 cm2 and below or equal 20 cm2 confirmed by the investigator's measurement, and its surface area not decreased by more than 40% compared to the selection value.

Exclusion Criteria

Patients who fulfill any of the following criteria are not eligible to be enrolled in the study:

1. Active Charcot foot, or inactive Charcot foot, if the target DFU cannot be properly offloaded.
2. Ulcers of non-neuropathic origin (e.g., rheumatoid, radiation-related, vasculitis-related ulcers).
3. Presence of any foot ulcer (whether or not on the target foot) for which local or systemic antibiotic treatment is required.
4. Evidence of skin cancer within or adjacent to the target ulcer.
5. Any infected ulcers, defined as any problem such as (but not limited to) cellulitis, osteomyelitis, gangrene, or deep tissue infection requiring local or systemic antibiotic therapy.
6. Another wound on the same foot as the target DFU. (i.e. Patients with another wound on the same limb as the target DFU are eligible for the study provided the concomitant wound is not infected and is above the ankle of the target foot).
7. Any known active malignancy that requires general, local, surgical or radiation therapy either ongoing or within the previous 6 months; or patients whose treatment has been suspended for compassionate reasons, or who are not considered as cured from any malignancy.
8. Morbid obesity, defined as body mass index (BMI) above or equal 45 kg/m2.
9. Clinically significant medical conditions, in the investigator's opinion, that could impair wound healing (e.g. hepatic impairment, immunocompromised patients).
10. Severe renal failure, defined as requirement for hemodialysis or peritoneal dialysis.
11. Females who are pregnant or breastfeeding, or who are of childbearing potential and not practicing a medically approved method of contraception.
12. Concomitant treatment with high dose oral or parenteral corticosteroids, defined as a daily dose of at least 7.5 mg prednisone or equivalent.
13. Participation in another clinical study within the previous 3 months.
14. Current participation in another clinical study with any drug or device.
15. History of drug or alcohol abuse within the previous year.
16. Concurrent severe psychiatric disease (including severe depressive disorder).
17. Known intolerance to the IMP or to any of its excipients.
18. Known to be uncooperative or noncompliant.
19. Outpatients who are unable to comply with the requirement for daily spray application at home (either application by a family member or by a visiting nurse).
20. Any other condition which, in the opinion of the investigator, would render the patient unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2010-12; Primary Completion 2012-05 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Charles Kerihuel, MD, Study Director — VERTICAL; Luc Téot, MD, Study Chair — Montpellier University Hospital
Locations (35):
- Belgium (3):
  - Brussels
  - Liège
  - Rumst
- Sofia, Bulgaria
- Croatia (3):
  - Crikvenica
  - Pula
  - Zagreb
- Aalborg, Denmark
- Germany (6):
  - Bad Mergentheim
  - Bad Nauheim
  - Cologne
  - Münster
  - Oldenburg
  - Trier
- Hungary (3):
  - LL, Budapest
  - PF, Budapest
  - Hatvan
- Netherlands (4):
  - Almelo
  - Amsterdam
  - Apeldoorn
  - Delft
- Poland (8):
  - Kalisz
  - Lodz
  - Lublin
  - Poznan
  - Szczecin
  - Warsaw
  - Wroclaw
  - Zielona Góra
- Slovakia (4):
  - Dunajská Streda
  - L'ubochna
  - Nové Zamky
  - Vráble
- Sweden (2):
  - EL, Malmo
  - ML, Malmo

RESULTS

PARTICIPANT FLOW:
Groups:
- Trafermin: Trafermin 0.01% spray: For ulcers with a maximum diameter (longest axis) of less or equal to 6 cm, the daily dose of trafermin 0.01% spray is 5 puffs (30 microgram) sprayed onto the wound surface. If the maximum diameter (longest axis) of the ulcer is >6 cm, the ulcer should be sprayed in two parts, i.e. 5 puffs (30 microgram) sprayed onto each half of the wound surface
- Placebo: Matching placebo spray: For ulcers with a maximum diameter (longest axis) of less or equal to 6 cm, the daily dose of trafermin 0.01% spray is 5 puffs (30 microgram) sprayed onto the wound surface. If the maximum diameter (longest axis) of the ulcer is >6 cm, the ulcer should be sprayed in two parts, i.e. 5 puffs (30 microgram) sprayed onto each half of the wound surface
Period: Overall Study
Arm/Group | Trafermin | Placebo
Started | 105 | 102
Completed | 93 | 95
Not Completed | 12 | 7
Not completed — Adverse Event | 6 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Surgery on the Target Limb | 0 | 2
Not completed — Protocol Deviation | 1 | 0
Not completed — Other | 2 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population was defined as all randomized patients who have at least one medical evaluation during the study. Demographic and baseline characteristics were presented in terms of descriptive statistics in ITT population.
Groups:
- Trafermin: Trafermin 0.01% spray
- Placebo: Matching placebo spray
- Total: Total of all reporting groups
Arm/Group | Trafermin | Placebo | Total
Number analyzed (Participants) | 105 | 102 | 207
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (9.0) | 59.4 (10.4) | 59.8 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 14 | 38
  Male | 81 | 88 | 169
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 104 | 102 | 206
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Wound size ≤5cm^2 [Number; unit: participants] | 81 | 80 | 161
Wound size >5cm^2 [Number; unit: participants] | 24 | 22 | 46
Peripheral blood perfusion Impaired [Number; unit: participants] | 17 | 16 | 33
Peripheral blood perfusion Normal [Number; unit: participants] | 88 | 86 | 174
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.19 (5.15) | 30.31 (4.92) | 30.25 (5.02)

OUTCOME MEASURES:

1. Primary Outcome: Wound Closure Rate of Diabetic Foot Ulcers (DFUs) of Neuropathic Origin After a Maximum of 12 Weeks Topical Daily Application of Trafermin 0.01% Spray Compared With Placebo, in Addition to Best Local Cares
Description: wound closure is defined as 100% reepithelialization of the target DFU, without exudates.
Time Frame: 12 weeks
Population: The primary analysis of the efficacy criteria was conducted on the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Trafermin | Placebo
Number analyzed (Participants) | 105 | 102
percentage of participants | 21.0 | 16.7
Statistical Analysis 1: Comparison: Trafermin vs Placebo; Test type: Superiority or Other; p = 0.4039, Regression, Logistic; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.66 to 2.80]

2. Secondary Outcome: Relative Wound Area Regression of 40% or More at 6 Week
Description: The incidence of wound area regression of at least 40% at week 6 was considered as an important exploratory secondary efficacy variable. The wound area regression was calculated as percentage change from inclusion at week 6 using centralized wound area data.
Time Frame: 6 weeks
Population: The analysis of the efficacy criteria was conducted on the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Trafermin | Placebo
Number analyzed (Participants) | 105 | 102
percentage of participants | 53.3 | 55.9
Statistical Analysis 1: Comparison: Trafermin vs Placebo; Test type: Superiority or Other; Regression, Logistic; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.52 to 1.56]

ADVERSE EVENTS:
Time Frame: Primary Treatment Emergent Adverse Event: adverse events that occurred after starting the treatment with the study medication until the end of primary follow up period up to 24 weeks.
Description: The safety population included all patients who were randomized and exposed to the study treatment.
Arm/Group | Trafermin | Placebo
Serious Adverse Events (participants affected / at risk) | 20/105 | 26/102
Other Adverse Events (participants affected / at risk) | 40/105 | 40/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trafermin (N=105) | Placebo (N=102)
Atrial fibrillation (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Sudden death (General disorders) | 0 | 1
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Diabetic foot infection (Infections and infestations) | 4 | 8
Erysipelas (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 1
Liver abscess (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 4
Pneumonia (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0
Glycosylated hemoglobin increased (Investigations) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 3 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Neuroglycopenia (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Transient ischemic attack (Nervous system disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Urinary tract inflammation (Renal and urinary disorders) | 0 | 1
Arteriovenous fistula (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Trafermin (N=105) | Placebo (N=102)
Edema peripheral (General disorders) | 7 | 11
Diabetic foot infection (Infections and infestations) | 9 | 12
Diabetic foot (Metabolism and nutrition disorders) | 24 | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI have no implicit or explicit rights to publish study data and results of their services.